CLINICAL TRIAL: NCT00769171
Title: A Prospective, Randomized, Double-blinded, Multi-center Trial Assessing the Safety and Efficacy of Intravenous Administration BAY12-8039 (Moxifloxacin) 400mg Every 24 h Compared to Intravenous Ceftriaxone 2g Every 24h and Metronidazole 500mg Every 12h for the Treatment of Patients With Complicated Intra-abdominal Infections
Brief Title: Dragon Study (the Safety and Efficacy for Treatment of Patients With Complicated Intra Abdominal Infections)
Acronym: DRAGON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11647
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Infection, Intra-abdominal
Keywords: Complicated Intra-Abdominal Infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — Moxifloxacin; Ceftriaxone; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Active Comparator)
  Interventions: Drug: Ceftriaxone + Metronidazole
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Moxifloxacin 400 mg every 24 h
  Arms: Arm 1
Drug: Ceftriaxone + Metronidazole — Ceftriaxone 2 g every 24 h and Metronidazole 500 mg every 12 h
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess the safety and efficacy of intravenous administration Moxifloxacin (BAY 12-8039) compared to intravenous ceftriaxone and metronidazole for the treatment of patients with complicated intra abdominal infections. In view of the fact that intra abdominal infections are typically polymicrobial and are often treated empirically, the selected antibacterial agent must cover the likely spectrum of bacterial pathogens. Combination antibiotics therapy has been widely used with great success.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized males or females >/= 18 years of age
* Expected duration of treatment with intravenous antibiotics in hospital is anticipated to be >/= 3 full days but not exceeding 14 days
* Ability to provide written informed consent
* Confirmed or suspected intra abdominal infection through surgical procedure or Radiological evidence. For suspected intra abdominal infection, The patient must be scheduled for a surgical procedure

Exclusion Criteria:

* Known hypersensitivity to fluoroquinolones, or other quinolones, and/or to beta lactams antibiotic drugs, or metronidazole or any of the excipients. History of tendon disease/disorder related to quinolone treatment
* Known congenital or documented acquired QT prolongation; uncorrected hypokalemia; clinically relevant bradycardia; clinically relevant heart failure with reduced left ventricular ejection fraction; previous history of symptomatic arrhythmias. Concomitant use of any of the following drugs, reported to increase the QT interval:
* Known severe end stage liver disease (Child Pugh C)
* Systemic antibacterial therapy for more than 24 h within 7 days of enrollment
* Indwelling peritoneal catheter, Pre existing ascites and presumed spontaneous bacterial peritonitis
* All pancreatic processes including pancreatic sepsis, peripancreatic sepsis, or an intra abdominal infection secondary to pancreatitis
* Traumatic perforation of the upper gastrointestinal tract (stomach, duodenum) or perforated peptic ulcer if duration of perforation is < 24 h or if operated on within 24 h of perforation
* Traumatic perforation of the small or large bowel if duration of perforation is < 12 h or if operated on within 12 h of perforation
* Transmural necrosis of the intestine due to acute embolic, thrombotic, or obstructive occlusions
* Acute cholecystitis with infection confined to the gallbladder unless there is evidence of an abscess or necrotic tissue or purulent exudate surrounding the gallbladder indicating a transition of bacteria and the inflammatory process into the abdominal cavity
* Early acute or suppurative, nonperforated appendicitis unless there is evidence of an abscess or peritoneal fluid containing leukocytes and micro organisms suggestive of regional contamination
* Infections originating from the female genital tract. Perinephric infections
* Severe, life threatening disease with a life expectancy of < 48 h or APS and APACHE scores of > 35, Known rapidly fatal underlying disease (death expected within 6 months)
* Neutropenia (neutrophil count < 1,000/microliter) caused by immunosuppressive therapy or malignancy
* Patients known to have AIDS or HIV seropositives who are receiving HAART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Clinical Response | After 10-14 days of treatment

SECONDARY OUTCOMES:
Clinical and bacteriological response | During 3-5days of treatment
Bacteriological and radiological response | After 10-14 days of treatment
Clinical response at the TOC visit in patients with bacteriological proven intra abdominal infection | After 10-14 days of treatment
Mortality attributable to intra abdominal infection | 13-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- China (6):
  - Nanjing, Jiangsu
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin
- Hong Kong (2):
  - Hong Kong, Hong Kong
  - Shatin, New Territories
- Bandung, West Java, Indonesia
- Malaysia (2):
  - Kuching, Sarawak
  - Terengganu
- South Korea (3):
  - Uijeongbu-si, Kyonggi-do
  - Incheon
  - Seoul
- Taiwan (3):
  - Tainan, Tainan
  - Kaoshiung
  - Taipei